CLINICAL TRIAL: NCT06047743
Title: Comparison of Upper and Lower Extremity Isometrics on Cognition in Healthy Adolescents: A Randomized Clinical Trial
Brief Title: Comparison of Upper and Lower Extremity Isometrics on Cognition in Healthy Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC-01640 Ramsha Abrar
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Healthy Adolescents
Keywords: Cognition; Isometrics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alternating unilateral Isometric Handgrip Exercise Group (Experimental): Participants (n=19) will be performing alternating unilateral Isometric Handgrip exercises using a dynamometer for 3-5 days a week for a total duration of 8 weeks. The participant will be seated with their elbow resting on the armrest and wrists off the supporting surface. A single session will consist of 4 sets of 30%MVC (calculated by dynamometer) of handgrip exercise with a maximum 2 minutes contraction time/ hold time followed by a rest period/ recovery period of 1 minute during each set.
  Interventions: Other: Alternating unilateral Isometric Handgrip Exercise
- Dominant knee extension Isometric Exercise Group (Experimental): Participants enrolled in this group will be performing dominant leg isometric knee extension. The knee will be 35° flexed from a fully extended position when performing isometric knee extension using a hand-held dynamometer retrained by a belt. The intervention duration will be 8 weeks. A single session will consist of performing 4 sets of 30% MVC (calculated using a dynamometer) of unilateral knee extension isometrics with a maximum 2 minutes contraction time/ hold time followed by a rest/ recovery period of 1 minute during each set.
  Interventions: Other: Dominant knee extension Isometric Exercise

INTERVENTIONS:
Other: Alternating unilateral Isometric Handgrip Exercise — Participants (n=19) will be performing alternating unilateral Isometric Handgrip exercises using a dynamometer for 3-5 days a week for a total duration of 8 weeks. The participant will be seated with their elbow resting on the armrest and wrists off the supporting surface. A single session will consist of 4 sets of 30%MVC (calculated by dynamometer) of handgrip exercise with a maximum 2 minutes contraction time/ hold time followed by a rest period/ recovery period of 1 minute during each set.
  Arms: Alternating unilateral Isometric Handgrip Exercise Group
Other: Dominant knee extension Isometric Exercise — Participants enrolled in this group will be performing dominant leg isometric knee extension. The knee will be 35° flexed from a fully extended position when performing isometric knee extension using a hand-held dynamometer retrained by a belt. The intervention duration will be 8 weeks. A single session will consist of performing 4 sets of 30% MVC (calculated using a dynamometer) of unilateral knee extension isometrics with a maximum 2 minutes contraction time/ hold time followed by a rest/ recovery period of 1 minute during each set.
  Arms: Dominant knee extension Isometric Exercise Group

SUMMARY:
This study aims to compare the effects of upper and lower-extremity isometrics on cognition in healthy adolescents.

DETAILED DESCRIPTION:
The literature suggests a positive impact of isometrics on cognition. Identifying how cognitive results would differ in upper vs. lower extremity isometric groups is the main objective of the study. for cognitive assessment, different aspects of cognition will be measured by all computer-based tools (except for Trail making A and B).

ELIGIBILITY:
Inclusion Criteria:

* School-going adolescents
* Both male and female students with a minimum age of 12 and a maximum of 18yrs
* Students with good school attendance
* Subjects who are willing to commit to the time commitments required by the program

Exclusion Criteria:

* Students with Physical or mental disabilities
* Those who suffered a fracture before
* Students with any morbidity

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Corsi Block Test | Baseline
  The Corsi block test or "Corsi block-tapping test" is a Short-term working memory (STM) task conceptually like the digital span test. Its creator is Philip Michael Corsi. In this test experimenter shows nine blocks arranged in front of the participant, The blocks are tapped in a certain sequence and the participant must repeat the same sequence. The test is repeated a few times with different lengths of blocks. The conclusion is drawn by observing the block/ corsi span. The block span is the longest sequence a participant can repeat. A healthy person has a block span of 5- 7.
Corsi Block Test | After 4 weeks
  The Corsi block test or "Corsi block-tapping test" is a Short-term working memory (STM) task conceptually like the digital span test. Its creator is Philip Michael Corsi. In this test experimenter shows nine blocks arranged in front of the participant, The blocks are tapped in a certain sequence and the participant must repeat the same sequence. The test is repeated a few times with different lengths of blocks. The conclusion is drawn by observing the block/ corsi span. The block span is the longest sequence a participant can repeat. A healthy person has a block span of 5- 7.
Corsi Block Test | After 8 weeks
  The Corsi block test or "Corsi block-tapping test" is a Short-term working memory (STM) task conceptually like the digital span test. Its creator is Philip Michael Corsi. In this test experimenter shows nine blocks arranged in front of the participant, The blocks are tapped in a certain sequence and the participant must repeat the same sequence. The test is repeated a few times with different lengths of blocks. The conclusion is drawn by observing the block/ corsi span. The block span is the longest sequence a participant can repeat. A healthy person has a block span of 5- 7.
Free and delayed recall test | Baseline
  Free and delayed recall are measures of episodic memory. A 15-item word list of highly frequent words will be used. At the outset, a "ready" cue will appear in the centre of the computer screen. On the computer screen, each word will be displayed individually for 3 seconds. After the 15th word, the participant will be given a 60-second to write down the words in any order. The Delayed Recall test will be used to evaluate long-term memory about 12 minutes later. During the delayed memory task, participants will be allowed 60 to recall as many words from the list shown before.
Free and delayed recall test | After 4 weeks
  Free and delayed recall are measures of episodic memory. A 15-item word list of highly frequent words will be used. At the outset, a "ready" cue will appear in the centre of the computer screen. On the computer screen, each word will be displayed individually for 3 seconds. After the 15th word, the participant will be given a 60-second to write down the words in any order. The Delayed Recall test will be used to evaluate long-term memory about 12 minutes later. During the delayed memory task, participants will be allowed 60 to recall as many words from the list shown before.
Free and delayed recall test | After 8 weeks
  Free and delayed recall are measures of episodic memory. A 15-item word list of highly frequent words will be used. At the outset, a "ready" cue will appear in the centre of the computer screen. On the computer screen, each word will be displayed individually for 3 seconds. After the 15th word, the participant will be given a 60-second to write down the words in any order. The Delayed Recall test will be used to evaluate long-term memory about 12 minutes later. During the delayed memory task, participants will be allowed 60 to recall as many words from the list shown before.
Go/ No Go task | Baseline
  Go/ No Go task or stop signal task is a measure of executive functioning. This tool tests participant's ability to not respond thus measuring response inhibition and impulsivity. The participant is required to respond within 2 seconds when the screen says 'Go' and should resist responding when 'No' appears.
Go/ No Go task | After 4 week
  Go/ No Go task or stop signal task is a measure of executive functioning. This tool tests participant's ability to not respond thus measuring response inhibition and impulsivity. The participant is required to respond within 2 seconds when the screen says 'Go' and should resist responding when 'No' appears
Go/ No Go task | After 8 weeks
  Go/ No Go task or stop signal task is a measure of executive functioning. This tool tests participant's ability to not respond thus measuring response inhibition and impulsivity. The participant is required to respond within 2 seconds when the screen says 'Go' and should resist responding when 'No' appears
Stroop test | Baseline
  The Stroop colour-word test is considered one of the gold standards of attentional measures and is one of the most widely used instruments in clinical and experimental neuropsychological settings. In the Stroop-A test, the reader must note the colour rather than the word as soon as the word is highlighted. In the Stroop-B, the evaluator points to the columns of coloured words, and the subject reads what is written. To draw results Stroop effect is calculated by subtracting the reaction time of compatible trials from incompatible trials.
Stroop test | After 4 weeks
  The Stroop colour-word test is considered one of the gold standards of attentional measures and is one of the most widely used instruments in clinical and experimental neuropsychological settings. In the Stroop-A test, the reader must note the colour rather than the word as soon as the word is highlighted. In the Stroop-B, the evaluator points to the columns of coloured words, and the subject reads what is written. To draw results Stroop effect is calculated by subtracting the reaction time of compatible trials from incompatible trials.
Stroop test | After 8 weeks
  The Stroop colour-word test is considered one of the gold standards of attentional measures and is one of the most widely used instruments in clinical and experimental neuropsychological settings. In the Stroop-A test, the reader must note the colour rather than the word as soon as the word is highlighted. In the Stroop-B, the evaluator points to the columns of coloured words, and the subject reads what is written. To draw results Stroop effect is calculated by subtracting the reaction time of compatible trials from incompatible trials.
Trail making A | Baseline
  The trail-making test is a cognitive tool used for the assessment of processing speed, attention, and cognitive flexibility. The test requires the person to draw lines in ascending order from 1-25 in the case of trail-making A. Trail-making A and B have numbers, as well as letters, joined in an alternating sequence. The total score is calculated by subtracting the time taken for part A from the time taken to attempt part B in seconds. If the person cannot complete the test in 5 minutes the test is discontinued.
Trail making B | Baseline
  The trail-making test is a cognitive tool used for the assessment of processing speed, attention, and cognitive flexibility. The test requires the person to draw lines in ascending order from 1-25 in the case of trail-making A. Trail-making A and B have numbers, as well as letters, joined in an alternating sequence. The total score is calculated by subtracting the time taken for part A from the time taken to attempt part B in seconds. If the person cannot complete the test in 5 minutes the test is discontinued.
Trail making A | After 4 weeks
  The trail-making test is a cognitive tool used for the assessment of processing speed, attention, and cognitive flexibility. The test requires the person to draw lines in ascending order from 1-25 in the case of trail-making A. Trail-making A and B have numbers, as well as letters, joined in an alternating sequence. The total score is calculated by subtracting the time taken for part A from the time taken to attempt part B in seconds. If the person cannot complete the test in 5 minutes the test is discontinued.
Trail making B | After 4 weeks
  The trail-making test is a cognitive tool used for the assessment of processing speed, attention, and cognitive flexibility. The test requires the person to draw lines in ascending order from 1-25 in the case of trail-making A. Trail-making A and B have numbers, as well as letters, joined in an alternating sequence. The total score is calculated by subtracting the time taken for part A from the time taken to attempt part B in seconds. If the person cannot complete the test in 5 minutes the test is discontinued.
Trail making A | After 8 weeks
  The trail-making test is a cognitive tool used for the assessment of processing speed, attention, and cognitive flexibility. The test requires the person to draw lines in ascending order from 1-25 in the case of trail-making A. Trail-making A and B have numbers, as well as letters, joined in alternating sequences. The total score is calculated by subtracting the time taken for part A from the time taken to attempt part B in seconds. If the person cannot complete the test in 5 minutes the test is discontinued.
Trail making B | After 8 weeks
  The trail-making test is a cognitive tool used for the assessment of processing speed, attention, and cognitive flexibility. The test requires the person to draw lines in ascending order from 1-25 in the case of trail-making A. Trail-making A and B have numbers, as well as letters, joined in alternating sequences. The total score is calculated by subtracting the time taken for part A from the time taken to attempt part B in seconds. If the person cannot complete the test in 5 minutes the test is discontinued.

SECONDARY OUTCOMES:
Borg Category-Ratio scale (CR)-10 Scale | Baseline
  The Borg Category-Ratio scale, also known as the Borg CR-10 scale, is a self-report tool for gauging perceived effort intensity. It is similar to the Borg Rating of Perceived Exertion Scale, but ratings are from 0 to 10. This general intensity scale has category-ratio qualities that are more suited to the subjective feelings of effort, including pain, discomfort, and localized tiredness. Participants will be cued to give their ratings using the standardized questions: "How hard do you feel your hand /leg muscles are working?" and will be scored against a rating of 0 to 10.
Borg Category-Ratio scale (CR)-10 Scale | After 4 weeks
  The Borg Category-Ratio scale, also known as the Borg CR-10 scale, is a self-report tool for gauging perceived effort intensity. It is similar to the Borg Rating of Perceived Exertion Scale, but ratings are from 0 to 10. This general intensity scale has category-ratio qualities that are more suited to the subjective feelings of effort, including pain, discomfort, and localized tiredness. Participants will be cued to give their ratings using the standardized questions: "How hard do you feel your hand /leg muscles are working?" and will be scored against a rating of 0 to 10.
Borg Category-Ratio scale (CR)-10 Scale | After 8 weeks
  The Borg Category-Ratio scale, also known as the Borg CR-10 scale, is a self-report tool for gauging perceived effort intensity. It is similar to the Borg Rating of Perceived Exertion Scale, but ratings are from 0 to 10. This general intensity scale has category-ratio qualities that are more suited to the subjective feelings of effort, including pain, discomfort, and localized tiredness. Participants will be cued to give their ratings using the standardized questions: "How hard do you feel your hand /leg muscles are working?" and will be scored against a rating of 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- Academy of Islamic and Modern Studies (AIMS), Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No